CLINICAL TRIAL: NCT01068743
Title: Bioequivalence Study of the Fixed Dose Combination of 2.5 mg Saxagliptin and 850 mg Metformin Tablet Relative to a 2.5 mg Saxagliptin (Onglyza) Tablet and a 850 mg Metformin (Glucophage Marketed by Merck Serono) Tablet Co-Administered to Healthy Subjects in the Fasted and Fed Conditions
Brief Title: Bioequivalence Study of Fixed Dose Combination of 2.5 mg Saxagliptin/850 mg Metformin Tablet Relative to 2.5 mg Onglyza and 850 mg Glucophage Tablets Co-Administered
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-121
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2012-02-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (saxagliptin 2.5 mg + metformin 850 mg; Fasting) (Other): A single oral dose of 2.5-mg Onglyza tablet and 850-mg Glucophage (marketed by Merck Serono) tablet administered together in the fasted condition.
  Interventions: Drug: saxagliptin; Drug: metformin
- Arm B (saxagliptin 2.5 mg + metformin 850 mg FDC; Fasting) (Other): A single oral dose of 2.5-mg saxagliptin/850-mg metformin fixed dose combination (FDC) administered in the fasted condition.
  Interventions: Drug: saxagliptin + metformin (FDC tablet)
- Arm C (saxagliptin 2.5 mg + metformin 850 mg; Fed) (Other): A single oral dose of 2.5-mg Onglyza tablet and 850-mg Glucophage (marketed by Merck Serono) tablet administered together in the fed condition.
  Interventions: Drug: saxagliptin; Drug: metformin
- Arm D (saxagliptin 2.5 mg + metformin 850 mg FDC; Fed) (Other): A single oral dose of 2.5-mg saxagliptin/850-mg metformin FDC administered in the fed condition.
  Interventions: Drug: saxagliptin + metformin (FDC tablet)

INTERVENTIONS:
Drug: saxagliptin — Tablets, Oral, 2.5 mg, once daily, single dose
  Other Names: Onglyza
  Arms: Arm A (saxagliptin 2.5 mg + metformin 850 mg; Fasting); Arm C (saxagliptin 2.5 mg + metformin 850 mg; Fed)
Drug: metformin — Tablets, Oral, 850 mg, once daily, single dose
  Other Names: Glucophage
  Arms: Arm A (saxagliptin 2.5 mg + metformin 850 mg; Fasting); Arm C (saxagliptin 2.5 mg + metformin 850 mg; Fed)
Drug: saxagliptin + metformin (FDC tablet) — Tablet, oral, (saxagliptin 2.5 mg) (metformin 850 mg), once daily, single dose
  Arms: Arm B (saxagliptin 2.5 mg + metformin 850 mg FDC; Fasting); Arm D (saxagliptin 2.5 mg + metformin 850 mg FDC; Fed)

SUMMARY:
To demonstrate bioequivalence of a 2.5 mg saxagliptin/850 mg metformin fixed dose combination (FDC) tablet relative to the 2.5 mg saxagliptin tablet and 850 mg metformin (Glucophage Marketed by Merck-Serono) tablet co-administered to healthy subjects in the fasted and fed condition.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 55 inclusive
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m^2, inclusive. BMI = weight (kg)/ [height (m)]^2

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* History of allergy to a dipeptidyl peptidase-IV (DPP4) inhibitor or related compound
* History of allergy or intolerance to metformin or other similar acting agents
* Prior exposure to saxagliptin
* Prior exposure to metformin within 3 months of study drug administration
* Estimated creatinine clearance (Clcr) of < 80 mL/min using the Cockcroft Gault formula

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (N = 24) who met all of the inclusion and none of the exclusion criteria were recruited from a single site in the United States.
Pre-assignment Details: Participants were screened for eligibility within 21 days before Day 1 of period 1. On Day -1 of each period, the participants were admitted to the clinical facility and confined for 4 days. All the 24 participants were randomly assigned to 1 of 4 treatment sequences (ADBC, BACD, CBDA, or DCAB). The washout between each dose was at least 7 days.
Groups:
- Treatment Sequence ADBC: Treatment A (period 1): 2.5 mg saxagliptin tablet + metformin 850 mg tablet single dose under fasted condition; Treatment D (period 2): Fixed dose combination (FDC) tablet (2.5 mg saxagliptin + metformin 850 mg) single dose under fed condition; Treatment B (period 3): FDC tablet (saxagliptin 2.5 mg + metformin 850 mg) single dose under fasted condition; Treatment C (period 4): 2.5 mg saxagliptin tablet + metformin 850 mg tablet single dose under fed condition.
- Treatment Sequence BACD: Treatment B (period 1): FDC tablet (saxagliptin 2.5 mg + metformin 850 mg) single dose under fasted condition; Treatment A (period 2): 2.5 mg saxagliptin tablet + metformin 850 mg tablet single dose under fasted condition; Treatment C (period 3): 2.5 mg saxagliptin tablet + metformin 850 mg tablet single dose under fed condition; Treatment D (period 4): Fixed dose combination (FDC) tablet (2.5 mg saxagliptin + metformin 850 mg) single dose under fed condition.
- Treatment Sequence CBDA: Treatment C (period 1): 2.5 mg saxagliptin tablet + metformin 850 mg tablet single dose under fed condition; Treatment B (period 2): FDC tablet (saxagliptin 2.5 mg + metformin 850 mg) single dose under fasted condition; Treatment D (period 3): Fixed dose combination (FDC) tablet (2.5 mg saxagliptin + metformin 850 mg) single dose under fed condition; Treatment A (period 4): 2.5 mg saxagliptin tablet + metformin 850 mg tablet single dose under fasted condition.
- Treatment Sequence DCAB: Treatment D (period 1): Fixed dose combination (FDC) tablet (2.5 mg saxagliptin + metformin 850 mg) single dose under fed condition; Treatment C (period 2): 2.5 mg saxagliptin tablet + metformin 850 mg tablet single dose under fed condition; Treatment A (period 3): 2.5 mg saxagliptin tablet + metformin 850 mg tablet single dose under fasted condition; Treatment B (period 4): FDC tablet (saxagliptin 2.5 mg + metformin 850 mg) single dose under fasted condition.
Period: Period 1
Arm/Group | Treatment Sequence ADBC | Treatment Sequence BACD | Treatment Sequence CBDA | Treatment Sequence DCAB
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence ADBC | Treatment Sequence BACD | Treatment Sequence CBDA | Treatment Sequence DCAB
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence ADBC | Treatment Sequence BACD | Treatment Sequence CBDA | Treatment Sequence DCAB
Started | 6 | 6 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Period 4
Arm/Group | Treatment Sequence ADBC | Treatment Sequence BACD | Treatment Sequence CBDA | Treatment Sequence DCAB
Started | 6 | 5 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled and Treated Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Height [Mean (Standard Deviation); unit: cm] | 170.2 (12.0)
Weight [Mean (Standard Deviation); unit: kg] | 79.7 (13.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (3.05)

OUTCOME MEASURES:

1. Primary Outcome: Saxagliptin Pharmacokinetic (PK) Parameter Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf])
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC (0-inf) is the area under the plasma concentration-time curve from time zero extrapolated to infinite time.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants not discontinuing prior to the end of the study. One participant in period 3 (treatment D) was excluded from the pharmacokinetic analysis due to a predose concentration greater than 5% of Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Treatment A: 2.5 mg saxagliptin tablet + metformin 850 mg tablet single dose under fasted condition
- Treatment B: Fixed dose combination (FDC) tablet (saxagliptin 2.5 mg + metformin 850 mg) single dose under fasted condition
- Treatment C: 2.5 mg saxagliptin tablet and metformin 850 mg tablet single dose under fed condition
- Treatment D: FDC tablet (2.5 mg saxagliptin + metformin 850 mg) single dose under fed condition
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 22
ng*hr/mL | 49.23 (18.52) | 49.94 (19.72) | 52.50 (17.95) | 53.15 (17.81)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; If there was no difference between the bioavailabilities of saxagliptin from the FDC tablet versus saxagliptin from coadministration of saxagliptin and metformin tablets under both fasted and fed conditions, then 20 participants would have provided 98% and 99% power to conclude bioequivalence (BE) with respect to Cmax and AUC0-inf, respectively. If there was a 5% difference, then 20 participants would have provided 93% and 99% power to conclude BE with respect to Cmax and AUC0-inf, respectively; Test type: Non-Inferiority or Equivalence — BE was concluded if the 90% confidence intervals (CIs) for the test-to-reference ratios (B/A) of geometric means were entirely contained within 80% to 125% for both Cmax and AUC0-inf of saxagliptin; Ratio (%) of Geometric LS Means = 101.45, 90% CI 2-sided [98.17 to 104.84] — Ratio=Treatment B/Treatment A. Geometric least squares means values are presented in other statistical analysis entries. LS=Least Squares
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; If there was no difference between the bioavailabilities of saxagliptin from the FDC tablet versus saxagliptin from coadministration of saxagliptin and metformin tablets under both fasted and fed conditions, then 20 participants would have provided 98% and 99% power to conclude BE with respect to Cmax and AUC0-inf, respectively. If there was a 5% difference, then 20 participants would have provided 93% and 99% power to conclude BE with respect to Cmax and AUC0-inf,respectively; Test type: Non-Inferiority or Equivalence — BE was concluded if the 90% CIs for the test-to-reference ratios (D/C) of geometric means were entirely contained within 80% to 125% for both Cmax and AUC0-inf of saxagliptin; Ratio (%) of Geometric LS Means = 102.43, 90% CI 2-sided [99.53 to 105.42] — Ratio=Treatment D/Treatment C. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 49.23
Statistical Analysis 4: Comparison: Treatment B; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 49.94
Statistical Analysis 5: Comparison: Treatment C; Geometric least squares means for Treatment C; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 52.71
Statistical Analysis 6: Comparison: Treatment D; Geometric least squares means for Treatment D; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 53.99

2. Secondary Outcome: 5-hydroxy Saxagliptin PK Parameter AUC(0-inf)
Description: as for outcome 1
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
ng*hr/mL | 118.58 (24.08) | 119.54 (21.16) | 121.99 (25.42) | 125.54 (24.82)

3. Secondary Outcome: 5-hydroxy Saxagliptin PK Parameter Cmax
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Cmax is the maximum observed concentration of drug substance in plasma.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
ng/mL | 16.83 (32.95) | 16.72 (32.92) | 17.35 (32.95) | 18.59 (30.78)

4. Primary Outcome: Saxagliptin PK Parameter Observed Maximum Plasma Concentration (Cmax)
Description: as for outcome 3
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 22
ng/mL | 9.73 (20.44) | 9.97 (29.07) | 10.25 (26.87) | 10.88 (23.72)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; If there was no difference between the bioavailabilities of saxagliptin from the FDC tablet versus saxagliptin from coadministration of saxagliptin and metformin tablets under both fasted and fed conditions, then 20 participants would have provided 98% and 99% power to conclude BE with respect to Cmax and AUC0-inf, respectively. If there was a 5% difference, then 20 participants would have provided 93% and 99% power to conclude BE with respect to Cmax and AUC0-inf, respectively; Test type: Non-Inferiority or Equivalence — BE was concluded if the 90% CIs for the test-to-reference ratios (B/A) of geometric means were entirely contained within 80% to 125% for both Cmax and AUC0-inf of saxagliptin; Ratio (%) of Geometric LS Means = 102.46, 90% CI 2-sided [94.68 to 110.88] — Ratio=Treatment B/Treatment A. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Ratio (%) of Geometric LS Means = 106.24, 90% CI 2-sided [98.43 to 114.66] — Ratio=Treatment D/Treatment C. Geometric least squares means values presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL) = 9.73
Statistical Analysis 4: Comparison: Treatment B; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL) = 9.97
Statistical Analysis 5: Comparison: Treatment C; Geometric least squares means for Treatment C; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL) = 10.33
Statistical Analysis 6: Comparison: Treatment D; Geometric least squares means for Treatment D; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL) = 10.97

5. Primary Outcome: Metformin PK Parameter AUC(0-inf)
Description: as for outcome 1
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 23 | 23 | 22
ng*hr/mL | 11998.00 (23.68) | 12271.61 (20.42) | 11988.30 (16.94) | 11838.11 (18.18)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; If there was no difference between the bioavailabilities of metformin from the FDC tablet versus metformin from coadministration of saxagliptin and metformin tablets under both fasted and fed conditions, then 20 participants would have provided 99% power to conclude BE with respect to each of Cmax and AUC0-inf. If there was a 5% difference, then 20 subjects would provide 97% and 99% power to conclude BE with respect to Cmax and AUC0-inf, respectively; Test type: Non-Inferiority or Equivalence — BE was concluded if the 90% CIs for the test-to-reference ratios (B/A) of geometric means were entirely contained within 80% to 125% for both Cmax and AUC0-inf of metformin; Ratio (%) of Geometric LS Means = 102.10, 90% CI 2-sided [97.26 to 107.18] — Ratio = Treatment B/Treatment A. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio (%) of Geometric LS Means = 99.17, 90% CI 2-sided [96.23 to 102.21] — Ratio=Treatment D/Treatment C. Geometric least squares means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares mean for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 11998
Statistical Analysis 4: Comparison: Treatment B; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 12250
Statistical Analysis 5: Comparison: Treatment C; Geometric least squares means for Treatment C; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 12036
Statistical Analysis 6: Comparison: Treatment D; Geometric least squares means for Treatment D; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 11937

6. Primary Outcome: Metformin PK Parameter Cmax
Description: as for outcome 3
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
ng/mL | 1724.38 (25.49) | 1715.79 (23.59) | 1571.21 (15.64) | 1541.76 (17.45)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Ratio (%) of Geometric LS Means = 99.50, 90% CI 2-sided [90.41 to 109.5] — Ratio=Treatment B/Treatment A. Geometric least squares means values presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — BE was concluded if the 90% CIs for the test-to-reference ratios (D/C) of geometric means were entirely contained within 80% to 125% for both Cmax and AUC0-inf of metformin; Ratio (%) of Geometric LS Means = 98.22, 90% CI 2-sided [94.28 to 102.32] — Ratio=Treatment D/Treatment C. Geometric least squares means values presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL = 1724.4
Statistical Analysis 4: Comparison: Treatment B; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Square Means (ng/mL) = 1715.8
Statistical Analysis 5: Comparison: Treatment C; Geometric least squares means for Treatment C; Test type: Superiority or Other; Geometric Least Square Mean (ng/mL) = 1581.4
Statistical Analysis 6: Comparison: Treatment D; Geometric least squares means for Treatment D; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL) = 1553.2

7. Secondary Outcome: 5-hydroxy Saxagliptin PK Parameter Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC[0-t])
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC[0-t] is the area under the plasma concentration-time curve from time zero to time of last measurable concentration.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
ng*hr/mL | 109.60 (25.81) | 110.61 (22.77) | 113.15 (26.53) | 117.04 (25.74)

8. Secondary Outcome: 5-hydroxy Saxagliptin PK Parameter Terminal Half-life (T 1/2)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. T 1/2 is the time required for the concentration of the drug to reach half of its original value in plasma.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
hr | 7.58 (1.32) | 7.58 (1.35) | 7.48 (1.10) | 7.22 (1.01)

9. Secondary Outcome: 5-hydroxy Saxagliptin PK Parameter Time to Achieve the Observed Maximum Plasma Concentration (Tmax)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Tmax is the time taken to reach the maximum observed plasma concentration.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
hr | 2.21 (0.75) | 1.86 (0.71) | 2.65 (0.83) | 2.46 (0.72)

10. Secondary Outcome: Safety: Adverse Events (AEs), Discontinuations Due to AEs, Deaths, and Serious AEs (SAEs).
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: AEs: from study drug administration Day 1/Period 1 till study discharge. SAEs: from date of written consent until 30 days after discontinuation of dosing or study participation. Duration of the study was approximately 45 days (including screening).
Population: All participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
participants
  Number of Participants With at Least 1 AE | 4 | 5 | 3 | 4
  Discontinuation Due to AE | 1 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0

11. Other Pre Specified Outcome: Saxagliptin PK Parameter AUC(0-t)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC(0-t) is the area under the plasma concentration-time curve from time zero to time of last measurable concentration.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 22
ng*hr/mL | 47.15 (17.98) | 47.83 (19.77) | 50.69 (17.74) | 51.37 (17.63)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; Ratio (%) of Geometric LS Means = 101.43, 90% CI 2-sided [98.07 to 104.90] — Ratio=Treatment B/Treatment A. Geometric least squares means values presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Superiority or Other; Ratio (%) of Geometric LS Means = 102.52, 90% CI 2-sided [99.56 to 105.57] — Ratio=Treatment D/Treatment C. Geometric least squares means values presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*h/mL) = 47.15 — Geometric least squares means for Treatment A
Statistical Analysis 4: Comparison: Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*h/mL) = 47.83 — Geometric least squares means for Treatment B
Statistical Analysis 5: Comparison: Treatment C; Test type: Superiority or Other; Geometric Least Squares Mean (ng*h/mL) = 50.89 — Geometric least squares means for Treatment C
Statistical Analysis 6: Comparison: Treatment D; Test type: Superiority or Other; Geometric Least Squares Mean (ng*h/mL) = 52.17 — Geometric least squares means for Treatment D

12. Other Pre Specified Outcome: Saxagliptin PK Parameter T1/2
Description: as for outcome 8
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 22
hr | 6.45 (1.00) | 6.21 (1.25) | 5.86 (0.92) | 6.09 (0.94)

13. Other Pre Specified Outcome: Saxagliptin PK Parameter Tmax
Description: as for outcome 9
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 22
hr | 1.38 (0.79) | 0.96 (0.61) | 1.94 (0.95) | 1.48 (0.58)

14. Other Pre Specified Outcome: Metformin PK Parameter AUC(0-t)
Description: as for outcome 11
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
ng*hr/mL | 11826.52 (23.86) | 11875.08 (21.47) | 11796.60 (17.03) | 11681.05 (17.59)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; Ratio (%) of Geometric LS Means = 100.41, 90% CI 2-sided [95.40 to 105.68] — Ratio=Treatment B/Treatment A. Geometric least squares means values presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Superiority or Other; Ratio (%) of Geometric LS Means = 99.06, 90% CI 2-sided [96.19 to 102.02] — Ratio=Treatment D/Treatment C. Geometric least squares means values presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*h/mL) = 11827 — Geometric least squares means for Treatment A
Statistical Analysis 4: Comparison: Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*h/mL) = 11875 — Geometric least squares means for Treatment B
Statistical Analysis 5: Comparison: Treatment C; Test type: Superiority or Other; Geometric Least Squares Mean (ng*h/mL) = 11845 — Geometric least squares means for Treatment C
Statistical Analysis 6: Comparison: Treatment D; Test type: Superiority or Other; Geometric Least Squares Mean (ng*h/mL) = 11734 — Geometric least squares means for Treatment D

15. Other Pre Specified Outcome: Metformin PK Parameter T1/2
Description: as for outcome 8
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 23 | 23 | 22
hr | 10.94 (4.13) | 13.15 (6.67) | 10.82 (3.18) | 11.13 (3.08)

16. Other Pre Specified Outcome: Metformin PK Parameter Tmax
Description: as for outcome 9
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
hr | 2.41 (0.78) | 2.54 (0.92) | 3.74 (0.54) | 3.74 (0.45)

17. Secondary Outcome: Safety: Clinically Significant Laboratory, Vital Sign, Physical Examination, and/or 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Abnormalities that were considered clinically significant and/or reported as an AE by the investigator.
Time Frame: From Day 1/Period 1 to study discharge or premature discontinuation. Duration of study was approximately 45 days (including screening).
Population: All participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 24 | 24 | 23 | 23
participants
  Clinical Laboratory Abnormalities | 0 | 0 | 1 | 0
  Vital Sign Abnormalities | 0 | 0 | 0 | 0
  Physical Examination Abnormalities | 0 | 0 | 0 | 0
  12-Lead ECG Abnormalities | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs: from study drug administration Day 1/Period 1 till study discharge. SAEs: from date of written consent until 30 days after discontinuation of dosing or study participation. Duration of the study was approximately 45 days (including screening).
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 4/24 | 5/24 | 3/23 | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=24) | Treatment B (N=24) | Treatment C (N=23) | Treatment D (N=23)
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1
Vessel puncture site pain (General disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period of <= 60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trail's primary publication.